CLINICAL TRIAL: NCT05317624
Title: Evaluation of Ultrasound Guided Platelet Rich Plasma Injection Versus Steroids Injection for Pain Relief in Cases of Partial Rotator Cuff Tears
Brief Title: Ultrasound Guided Steroids Injection Versus PRP for Shoulder Pain Relief
Acronym: PRP
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, radwa saber, Radwa saber, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0201491
Record Dates: First submitted 2021-07-19; First posted 2022-04-08 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2022-09

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain | interventions — Methylprednisolone

STUDY DESIGN:
Intervention Model Description: 2 groups will be included
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Platelet rich plasma group (Experimental): participants will receive Ultrasound guided subacromial injection of 3 ml platelet rich plasma+0.5 ml of PRP activator (10% calcium gluconate)+ 1ml 0.5%bupivacaine.
  Interventions: Combination Product: Platelet rich plasma
- Methylprednisolone group (Experimental): participants will receive Ultrasound guided subacromial injection of 1 ml methylprednisolone+ 1ml 0.5%bupivacaine + 2.5 ml normal saline.
  Interventions: Combination Product: Methylprednisolone

INTERVENTIONS:
Combination Product: Platelet rich plasma — platelet rich plasma will be obtained from the particepants own blood mixed with activator and bupivacaine
  Other Names: PRP group
  Arms: Platelet rich plasma group
Combination Product: Methylprednisolone — 1ml methyl prednisolone 40mg\ml mixed with normal saline and bupivacaine
  Other Names: steroids group
  Arms: Methylprednisolone group

SUMMARY:
Comparison between effects of ultrasound guided platelet rich plasma injection versus steroids injection for pain relief in cases of partial rotator cuff tears

DETAILED DESCRIPTION:
The effect of injection of platelet rich plasma will be compared with effects of steroids injection according to pain relief effects,, Side effects ,, healing ability ,, recurrence in both groups.

30 patient in each group will be included

ELIGIBILITY:
Inclusion Criteria:

1. Patients with positive tests for rotator cuff pain
2. Patients with positive radiological (US or MRI) findings of partial rotator cuff tear

Exclusion Criteria:

1. Patient refusal
2. Age less than 20 years.
3. Infection at injection site.
4. Prior surgery on the shoulder joint area.
5. Presence of other associated pathology in the shoulder joint
6. Patients using antiplatelet drugs (aspirin).
7. Contraindications to the use of platelet concentrate
8. Contraindications to the steroids injection

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Shoulder pain assesment | 4 months
  The pain will be assessed using visual analogue scale( score range=0-10,less than 4,4-6 and more than 6 for mild, moderate and severe pain respectively)

SECONDARY OUTCOMES:
Assesment of rotator cuff tendon healing | 4 months
  assesment healing process of tendon using ultrasound technique
Assesment the failure rate after shoulder joint injection | 4 months
  failure of relief the symptoms after shoulder joint injection will be recorded
The reinjection rate recording | 4 months
  the incidence of reinjection the shoulder joint due to inadequate pain relief will be recorded
Assesment the rate of tear recurrence after shoulder joint injection | 4 months
  The rate of tear recurrence after 4 months of injection will be assessed using MRI or US
Simple shoulder assessment test | 4 months
  Functional assessment of shoulder joint will be done using simple sholder assessment test 0= maximal disability 20% -40% = crippled 40% -60% = severe disability 60% -80% = moderate disability 100% = no disability

OTHER OUTCOMES:
Measurement plasma C-Reactive Protein level | 4 months
  The plasma C- Reactive Protein level will be measured prior to injection and 4 months later on after the procedure
Measurement the fasting blood glucose level | one week
  The fasting blood glucose level will be measure prior to and one week later after injection
Assesment the complications after shoulder joint injection | 4 months
  Complications that might occur after shoulder joint injection such as infection, elevated blood sugar, allergy, nerve injury, nausea and vomiting will be recorded
Measurement the serum cortisol level | one week
  Early morning(8 am serum cortisol level) will be measured before the injection and one week later after injection

CONTACTS AND LOCATIONS:
Overall Officials: Dorreya Fikry, Principal Investigator — AlexandriaUniversity; Tarek Sarhan, Study Director — AlexandriaUniversity
Locations (1):
- Facility of medicine, Alexandria, Egypt